CLINICAL TRIAL: NCT00136305
Title: Relative Effectiveness of Pictorial and Written Asthma Action Plans for Pediatric Asthma
Brief Title: Comparing Asthma Action Plans for Pediatric Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI moved to a different institution
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Katherine B. Anderson Associates Endowment Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04 08-102E; KBR 01.4182
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Asthma
Keywords: pediatric asthma; asthma action plans; patient education; medication adherence
MeSH Terms: conditions — Asthma; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pictorial Asthma Action Plan (Experimental)
  Interventions: Behavioral: Pictorial asthma action plan
- Written Asthma Action Plan (Active Comparator)
  Interventions: Behavioral: Written asthma action plan

INTERVENTIONS:
Behavioral: Pictorial asthma action plan
  Arms: Pictorial Asthma Action Plan
Behavioral: Written asthma action plan
  Arms: Written Asthma Action Plan

SUMMARY:
The purpose of this study is to evaluate and compare the relative effectiveness of two asthma action plans (pictorial versus written) in terms of asthma action plan knowledge, medication use, and family satisfaction with asthma education.

DETAILED DESCRIPTION:
Asthma medical regimens are complex for families, requiring changes in the types and amounts of medication based on the frequency and intensity of symptoms. Written asthma action plans (AAP's) are commonly used to provide a set of instructions to help parents and children implement these complicated regimens. However, written AAP's require substantial literacy levels, so for younger children, low-literacy families, or non-English speaking families, a pictorial version of the AAP may be more understandable and useful. The study aims to validate a newly developed, fully pictorial AAP in terms of its relative impact on parent- and child-reported knowledge of the action plan, medication use, and parent- and child-reported satisfaction, when compared to a standard-care written AAP.

ELIGIBILITY:
Inclusion Criteria:

* Children who are new patients
* Receive a diagnosis of persistent asthma
* Are in need of an asthma action plan

Exclusion Criteria:

* Diagnosed with intermittent asthma
* An established patient who already has an asthma action plan
* Not English or Spanish speaking

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2005-08; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Scores on the Asthma Action Plan Knowledge Interview | 1 month
  Measures recall of asthma treatment plan

SECONDARY OUTCOMES:
Adherence to Controller Medication | 1 month
  Mean daily adherence to medication measured via electronic monitoring
Rescue Medication Use | 1 month
  Number of puffs of inhaled rescue medication
Family satisfaction survey scores | 1 month
  Family ratings of satisfaction with asthma action plan

CONTACTS AND LOCATIONS:
Overall Officials: Christina D Adams, PhD, Principal Investigator — The Children's Mercy Hospitals and Clinics
Locations (1):
- The Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States